CLINICAL TRIAL: NCT04278924
Title: A Phase 2, Randomized, Double-blind, Placebo-Controlled Study to Evaluate Safety, Tolerability, and Efficacy of TAK-079 in Patients With Persistent/Chronic Primary Immune Thrombocytopenia
Brief Title: A Study of TAK-079 in Adults With Persistent/Chronic Primary Immune Thrombocytopenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-079-1004; 2019-004103-12 (EudraCT Number); jRCT2031220408 (Registry Identifier: jRCT)
Record Dates: First submitted 2020-02-19; First posted 2020-02-20 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: Drug Therapy
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A & B: Double Blind Period: Placebo (Placebo Comparator): Participants received TAK-079 placebo-matching injection subcutaneously (SC), once weekly (QW) for 8 weeks. Following treatment participants were followed up for 8 weeks in a double blinded short follow-up period (SFP) up to Week 16. Participants who opted to receive treatment with TAK-079 were then randomized to receive TAK-079, SC injection, QW for 8 weeks in Open-label Extension (OLE) Period of Part A or Part B. Participants who did not opt to receive treatment with TAK-079 were followed up for another 16 weeks in an unblinded long follow-up period (LFP) up to Week 32.
  Interventions: Drug: Placebo
- Part A: Double Blind Period: TAK-079 100 mg (Experimental): Participants received TAK-079 100 mg, SC injection, QW for 8 weeks. Following treatment participants were followed up for 8 weeks in a double blinded SFP up to Week 16. Participants who opted to receive treatment with TAK-079 were then randomized to receive TAK-079, SC injection, QW for 8 weeks in OLE Period of Part A or Part B. Participants who did not opt to receive treatment with TAK-079 were followed up for another 16 weeks in an unblinded LFP up to Week 32.
  Interventions: Drug: TAK-079
- Part A: Double Blind Period: TAK-079 300 mg (Experimental): Participants received TAK-079 300 mg, SC injection, QW for 8 weeks. Following treatment participants were followed up for 8 weeks in a double blinded SFP up to Week 16. Participants who opted to receive treatment with TAK-079 were then randomized to receive TAK-079, SC injection, QW for 8 weeks in OLE Period of Part A or Part B. Participants who did not opt to receive treatment with TAK-079 were followed up for another 16 weeks in an unblinded LFP up to Week 32.
  Interventions: Drug: TAK-079
- Part B: Double Blind Period: TAK-079 600 mg (Experimental): Participants received TAK-079 600 mg, SC injection, QW for 8 weeks. Following treatment participants were followed up for 8 weeks in a double blinded SFP up to Week 16. Participants who opted to receive treatment with TAK-079 were then randomized to receive TAK-079, SC injection, QW for 8 weeks in OLE Period of Part A or Part B. Participants who did not opt to receive treatment with TAK-079 were followed up for another 16 weeks in an unblinded LFP up to Week 32.
  Interventions: Drug: TAK-079
- Part A: Open-label Extension (OLE) Period: TAK-079 100 mg (Experimental): Participants who received placebo in double-blind Part A and opted to receive treatment with TAK-079 were randomized to receive TAK-079 100 mg, SC injection, QW for 8 weeks in OLE Period of Part A. Following treatment participants were followed up for 8 weeks in a SFP and then for another 16 weeks in a LFP.
  Interventions: Drug: TAK-079
- Part A: OLE Period: TAK-079 300 mg (Experimental): Participants who received placebo in double-blind Part A and opted to receive treatment with TAK-079 were randomized to receive TAK-079 300 mg, SC injection, QW for 8 weeks in OLE Period of Part A. Following treatment participants were followed up for 8 weeks in a SFP and then for another 16 weeks in a LFP.
  Interventions: Drug: TAK-079
- Part B: OLE Period: TAK-079 600 mg (Experimental): Participants who received placebo in double-blind Part B and opted to receive treatment with TAK-079 received TAK-079 600 mg, SC injection, QW for 8 weeks in OLE Period of Part B. Following treatment participants were followed up for 8 weeks in a SFP and then for another 16 weeks in a LFP.
  Interventions: Drug: TAK-079

INTERVENTIONS:
Drug: Placebo — TAK-079 placebo-matching SC injection.
  Arms: Part A & B: Double Blind Period: Placebo
Drug: TAK-079 — TAK-079 SC injection.
  Arms: Part A: Double Blind Period: TAK-079 100 mg; Part A: Double Blind Period: TAK-079 300 mg; Part A: OLE Period: TAK-079 300 mg; Part A: Open-label Extension (OLE) Period: TAK-079 100 mg; Part B: Double Blind Period: TAK-079 600 mg; Part B: OLE Period: TAK-079 600 mg

SUMMARY:
Primary immune thrombocytopenia (ITP) is a rare disease that results in low levels of platelets - the cells that help blood clot.

The main aim of the study is to check for side effects from taking TAK-079 at three different dose levels. Another aim is to learn if TAK-079 can increase the platelet count in people with ITP.

In addition to receiving stable background therapy for ITP, participants will receive an injection of either TAK-079 or a placebo once a week for 2 months. A placebo looks like TAK-079 but will not have any medicine in it. After treatment, all participants will be followed-up for another 2 months.

Then, participants who received TAK-079 will continue to be followed-up for an extra 4 months. Participants who received the placebo and would like to receive TAK-079 may be able to do this in an extension period in the study.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-079. TAK-079 is being tested to treat people who have primary immune thrombocytopenia (ITP). This study will evaluate the safety and biologic activity of TAK-079 or matching placebo in combination with stable ITP background therapy.

The study will enroll approximately 36 to 54 participants. In Part A of the study, participants will be randomly assigned (by chance, like flipping a coin) to one of the three treatment groups. Those who received placebo in this period will have the choice to receive TAK-079 after a safety follow-up period and will be randomized to one of the two open-label TAK-079 treatment arms. An unblinded safety review will take place once a minimum of 24 evaluable participants are available for analysis in Part A to decide whether to open enrollment into Part B.

In Part B participants will be randomly assigned to one of two treatment groups. Those who received placebo in this period will have the choice to receive study drug after a safety follow-up period in a single open-label TAK-079 treatment arm.

This multi-center trial will be conducted worldwide. All participants will be followed for at least 8 weeks in a Safety Follow-up Period, and a 16-week Long-term Follow-up Period after the 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with ITP that has persisted for ≥3 months, diagnosed in accordance to The American Society of Hematology 2011 Evidence-based Practice Guideline for Immune Thrombocytopenia or the International Consensus Report on The Investigation and Management of Primary Immune Thrombocytopenia as locally applicable.
2. Has a mean platelet count of <30,000/μL (and individually ≤35,000/μL) on at least 2 measurements at least 1 week apart during screening.
3. Diagnosis of ITP supported by a prior response to an ITP therapy (other than a thrombopoietin receptor agonists [TPO-RA]) that achieved a platelet count of ≥50,000/μL.
4. If receiving standard background treatment for ITP, treatment should be stable in dose and frequency for at least 4 weeks before dosing.

   1. Permitted standard background treatments may include: 1 oral corticosteroid; ±1 immunosuppressant from the following list: azathioprine, danazol, dapsone, cyclosporine, mycophenolate mofetil, mycophenolate sodium; ±1 TPO-RA (romiplostim, eltrombopag, avatrombopag); ±fostamatinib. Corticosteroids, including dexamethasone, must be given as oral, daily or every-other-day therapy as opposed to pulse therapy.
   2. The dose of any permitted standard background therapy must be expected to remain stable through the study, unless dose reduction is required because of toxicities.

Exclusion Criteria:

1. Use of anticoagulants or any drug with antiplatelet effect (such as aspirin) within 3 weeks before screening.
2. Has a history of any thrombotic or embolic event within 12 months before screening.
3. Has a history of splenectomy within 3 months before screening.
4. Use of intravenous immunoglobulin (IVIg), subcutaneous immunoglobulin or anti-D immunoglobulin treatment within 4 weeks of screening, or an expectation that any therapy besides the participant's standard background therapies may be used for treatment of thrombocytopenia (e.g., a rescue therapy) between screening and dosing.
5. Diagnosed with chronic obstructive pulmonary disease (COPD) or asthma, and a prebronchodilatory forced expiratory volume in 1 second (FEV1) <50% of predicted normal.
6. Use of rituximab or any monoclonal antibody (mAb) for immunomodulation within 4 months before first dosing. Note: Participants with prior exposure to rituximab must have cluster of differentiation (CD) 19 counts within the normal range at screening.
7. Use of immunosuppressants (such as cyclophosphamide, vincristine) other than permitted oral immunosuppressants within 6 months before first dosing.
8. Has been diagnosed with myelodysplastic syndrome.
9. Has received a live vaccine within 4 weeks before screening or has any live vaccine planned during the study.

10 Has had an opportunistic infection ≤12 weeks before initial study dosing or is currently undergoing treatment for a chronic opportunistic infection, such as tuberculosis (TB), pneumocystis pneumonia, cytomegalovirus, herpes simplex virus, herpes zoster, or atypical mycobacteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (55):
- United States (7):
  - Arizona Clinical Research Center - Hunt - PPDS, Tucson, Arizona
  - University of Florida, Gainesville, Florida
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Leo W. Jenkins Cancer Center, Greenville, North Carolina
  - University of Virginia, Charlottesville, Virginia
- Bulgaria (6):
  - Acibadem City Clinic Multiprofile Hospital for Active Treatment Tokuda, Sofia, Sofia-Grad
  - University Multiprofile Hospital for Active Treatment Sofiamed OOD, Sofia, Sofia-Grad
  - University Multiprofile Hospital for Active Treatment - Dr. Georgi Stranski EAD, Pleven
  - University Mulitiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - University Multiprofile Hospital for Active Treatment Sv Ivan Rilski EAD, Sofia
  - Military Medical Academy Multiprofile Hospital for Active Treatment - Sofia, Sofia
- China (2):
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
- Croatia (3):
  - Clinical Hospital Centre Osijek, Osijek
  - Klinicki bolnicki centar Zagreb, Zagreb
  - University Hospital Merkur, Zagreb
- Germany (4):
  - Universitatsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Onkologische Schwerpunktpraxis Kurfurstendamm, Berlin
  - OnkoNet Marburg GmbH, Marburg
  - Rotkreuzklinikum Munchen, München
- Greece (3):
  - University General Hospital of Patras, Pátrai, Achaia
  - General Hospital of Athens - George Gennimatas, Athens, Attica
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Italy (7):
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI), Trieste, Friuli Venezia Giulia
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Azienda Ospedaliera Di Rilievo Nazionale E Di Alta Specializzazione Garibaldi, Catania, Sicily
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - A.O.U. Maggiore della Carita, Novara
  - Azienda Policlinico Umberto I, Roma
- Japan (2):
  - Saiseikai Central Hospital, Minato-Ku, Tokyo
  - Nihon University Itabashi Hospital, tabashi City, Tokyo
- Slovenia (2):
  - Univerzitetni klinicni Center Ljubljana, Ljubljana
  - University Clinical Centre Maribor, Maribor
- Spain (12):
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Principe de Asturias, Meco, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital del Mar, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - C.A.U de Burgos - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Quironsalud Madrid, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Málaga
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Ukraine (7):
  - Municipal Non-profit Enterprise Mykolayiv Regional Clinical Hospital the Mykolayiv Regional Council, Mykolaiv, Mykolaivs'ka Oblast
  - Municipal Non-profit Enterprise Ternopil Regional Clinical Hospital of Ternopil Regional Council, Ternopil, Ternopil Oblast
  - MNE Regional Clinical Hospital n a O F Herbachevskyi of Zhytomyr Regional Council, Zhytomyr, Zhytomyr Oblast
  - Municipal Non-profit Enterprise "City Clinical Hospital # 4" of Dnipro City Council - PPDS, Dnipro
  - Medical Center OK!Clinic+LLC International Institute of Clinical Research, Kyiv
  - CNE Kyiv City Clinical Hospital #9 of Exec. Body of Kyiv City Council Kyiv City State Admin, Kyiv
  - State Institution Institute of Blood Pathology and Transfusion Medicine of NAMS of Ukraine, Lviv

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b603d4db2bf003ab4a391?idFilter=%5B%22TAK-079-1004%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 24 investigative sites globally from 09 November 2020 to 29 April 2024.
Pre-assignment Details: Participants who had persistent/chronic primary immune thrombocytopenia (ITP) were randomized to receive either mezagitamab (TAK-079) or matching placebo in Part A or Part B of this study.
Groups:
- Part A & B: Double Blind Period: Placebo: Participants received TAK-079 placebo-matching injection subcutaneously (SC), once weekly (QW) for 8 weeks. Following treatment participants were followed up for 8 weeks in a double blinded short follow-up period (SFP) up to Week 16. Placebo-assigned participants who did not opt to receive treatment with TAK-079 were followed up for another 16 weeks in an unblinded long follow-up period (LFP) up to Week 32.
- Part A: Double Blind Period: TAK-079 100 mg: Participants received TAK-079 100 mg, SC injection, QW for 8 weeks. Following treatment participants were followed up for 8 weeks in a double blinded SFP up to Week 16. Participants were then followed up for another 16 weeks in an unblinded LFP up to Week 32.
- Part A: Double Blind Period: TAK-079 300 mg: Participants received TAK-079 300 mg, SC injection, QW for 8 weeks. Following treatment participants were followed up for 8 weeks in a double blinded SFP up to Week 16. Participants were then followed up for another 16 weeks in an unblinded LFP up to Week 32.
- Part B: Double Blind Period: TAK-079 600 mg: Participants received TAK-079 600 mg, SC injection, QW for 8 weeks. Following treatment participants were followed up for 8 weeks in a double blinded SFP up to Week 16. Participants were then followed up for another 16 weeks in an unblinded LFP up to Week 32.
Period: Double Blind Period (Main Study)
Arm/Group | Part A & B: Double Blind Period: Placebo | Part A: Double Blind Period: TAK-079 100 mg | Part A: Double Blind Period: TAK-079 300 mg | Part B: Double Blind Period: TAK-079 600 mg | Part A: Open-label Extension (OLE) Period: TAK-079 100 mg | Part A: OLE Period: TAK-079 300 mg | Part B: OLE Period: TAK-079 600 mg
Started | 13 | 9 | 8 | 11 | 0 | 0 | 0
Completed | 12 | 7 | 8 | 9 | 0 | 0 | 0
Not Completed | 1 | 2 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Open-label Extension Period
Arm/Group | Part A & B: Double Blind Period: Placebo | Part A: Double Blind Period: TAK-079 100 mg | Part A: Double Blind Period: TAK-079 300 mg | Part B: Double Blind Period: TAK-079 600 mg | Part A: Open-label Extension (OLE) Period: TAK-079 100 mg | Part A: OLE Period: TAK-079 300 mg | Part B: OLE Period: TAK-079 600 mg
Started | 0 | 0 | 0 | 0 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Part A & B: Double Blind Period: Placebo: Participants received TAK-079 placebo-matching injection SC, QW for 8 weeks. Following treatment participants were followed up for 8 weeks in a double blinded SFP up to Week 16. Placebo-assigned participants who did not opt to receive treatment with TAK-079 were followed up for another 16 weeks in an unblinded LFP up to Week 32.
- Total: Total of all reporting groups
Arm/Group | Part A & B: Double Blind Period: Placebo | Part A: Double Blind Period: TAK-079 100 mg | Part A: Double Blind Period: TAK-079 300 mg | Part B: Double Blind Period: TAK-079 600 mg | Total
Number analyzed (Participants) | 13 | 9 | 8 | 11 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (15.86) | 49.0 (14.45) | 52.3 (16.59) | 48.4 (19.68) | 46.2 (17.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 5 | 9 | 28
  Male | 4 | 4 | 3 | 2 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 12 | 9 | 8 | 9 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 11 | 9 | 8 | 9 | 37
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Grade 3 or Higher Treatment Emergent Adverse Event (TEAE), Treatment Emergent Serious Adverse Event (SAE), and TEAEs Leading to TAK-079 Discontinuation
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with the treatment. SAE means any untoward medical occurrence that at any dose: a) results in death; b) is life-threatening; c) requires inpatient hospitalization or prolongation of an existing hospitalization; d) results in persistent or significant disability or incapacity; e) is a congenital anomaly/birth defect; f) is a medically important event. TEAEs were defined as an AE having a start date and time equal to or later than the start date and time of the first dose of investigational medicinal product (IMP). Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to Week 32 in each Period of the study
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A & B: Double Blind Period: Placebo | Part A: Double Blind Period: TAK-079 100 mg | Part A: Double Blind Period: TAK-079 300 mg | Part B: Double Blind Period: TAK-079 600 mg | Part A: Open-label Extension (OLE) Period: TAK-079 100 mg | Part A: OLE Period: TAK-079 300 mg | Part B: OLE Period: TAK-079 600 mg
Number analyzed (Participants) | 13 | 9 | 8 | 11 | 4 | 4 | 4
percentage of participants
  Grade 3 or Higher TEAE | 23.1 | 22.2 | 0 | 27.3 | 0 | 0 | 25.0
  Treatment Emergent SAE | 7.7 | 22.2 | 0 | 18.2 | 25.0 | 0 | 0
  TEAEs Leading to TAK-079 Discontinuation | 0 | 22.2 | 0 | 18.2 | 25.0 | 0 | 0

2. Secondary Outcome: Percentage of Participants With Platelet Response at Weeks 16 and 32
Description: Platelet response is defined as a platelet count ≥50,000/microliter (μL) and ≥20,000/μL above baseline on at least 2 visits without a dosing period-permitted rescue treatment in the previous 4 weeks and without any other previous rescue therapy. Percentages were rounded off to the nearest single decimal place.
Time Frame: At Weeks 16 and 32
Population: The Full Analysis Set included all randomized participants who had received at least 1 dose of study drug. Number analyzed indicates the number of participants with data available for analyses at the specified time point. All participants in the 'Part A & B: Double Blind Period: Placebo' arm either transitioned to OLE Period or discontinued from the study prior to Week 32.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A & B: Double Blind Period: Placebo | Part A: Double Blind Period: TAK-079 100 mg | Part A: Double Blind Period: TAK-079 300 mg | Part B: Double Blind Period: TAK-079 600 mg | Part A: Open-label Extension (OLE) Period: TAK-079 100 mg | Part A: OLE Period: TAK-079 300 mg | Part B: OLE Period: TAK-079 600 mg
Number analyzed (Participants) | 13 | 9 | 8 | 11 | 4 | 4 | 4
percentage of participants
  Week 16 | 23.08 [5.04 to 53.81] | 66.67 [29.93 to 92.51] | 62.50 [24.49 to 91.48] | 90.91 [58.72 to 99.77] | 50.00 [6.76 to 93.24] | 50.00 [6.76 to 93.24] | 25.00 [0.63 to 80.59]
  Week 32: number analyzed (Participants) | 0 | 9 | 8 | 11 | 4 | 4 | 4
  Week 32 |  | 66.67 [29.93 to 92.51] | 62.50 [24.49 to 91.48] | 90.91 [58.72 to 99.77] | 50.00 [6.76 to 93.24] | 50.00 [6.76 to 93.24] | 25.00 [0.63 to 80.59]
Statistical Analysis 1: Comparison: Part A & B: Double Blind Period: Placebo vs Part A: Double Blind Period: TAK-079 100 mg; Test type: Superiority; p = 0.056, Barnard's test; Risk Difference (RD) = 43.59, 95% CI 2-sided [0.81 to 73.35] — 95% confidence interval (CI) of the difference in percentage was calculated using Miettinen-Nurminen method
Statistical Analysis 2: Comparison: Part A & B: Double Blind Period: Placebo vs Part A: Double Blind Period: TAK-079 300 mg; Test type: Superiority; p = 0.088, Barnard's test; Risk Difference (RD) = 39.42, 95% CI 2-sided [-4.24 to 71.38] — 95% CI of the difference in percentage was calculated using Miettinen-Nurminen method
Statistical Analysis 3: Comparison: Part A & B: Double Blind Period: Placebo vs Part B: Double Blind Period: TAK-079 600 mg; Test type: Superiority; p = 0.001, Barnard's test; Risk Difference (RD) = 67.83, 95% CI 2-sided [29.21 to 87.29] — 95% CI of the difference in percentage was calculated using Miettinen-Nurminen method

3. Secondary Outcome: Percentage of Participants With Complete Platelet Response at Weeks 16 and 32
Description: Complete platelet response is defined as a platelet count ≥100,000/μL on at least 2 visits without a dosing period-permitted rescue treatment in the previous 4 weeks and without any other previous rescue therapy. Percentages were rounded off to the nearest single decimal place.
Time Frame: At Weeks 16 and 32
Population: The Full Analysis Set consisted of all randomized participants who had received at least 1 dose of study drug. Number analyzed indicates the number of participants with data available for analyses at the specified time point. All participants in the 'Part A & B: Double Blind Period: Placebo' arm either transitioned to OLE Period or discontinued from the study prior to Week 32.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A & B: Double Blind Period: Placebo | Part A: Double Blind Period: TAK-079 100 mg | Part A: Double Blind Period: TAK-079 300 mg | Part B: Double Blind Period: TAK-079 600 mg | Part A: Open-label Extension (OLE) Period: TAK-079 100 mg | Part A: OLE Period: TAK-079 300 mg | Part B: OLE Period: TAK-079 600 mg
Number analyzed (Participants) | 13 | 9 | 8 | 11 | 4 | 4 | 4
percentage of participants
  Week 16 | 0 [0.00 to 24.71] | 55.56 [21.20 to 86.30] | 50.00 [15.70 to 84.30] | 81.82 [48.22 to 97.72] | 0 [0.00 to 60.24] | 25.00 [0.63 to 80.59] | 25.00 [0.63 to 80.59]
  Week 32: number analyzed (Participants) | 0 | 9 | 8 | 11 | 4 | 4 | 4
  Week 32 |  | 55.56 [21.20 to 86.30] | 50.00 [15.70 to 84.30] | 81.82 [48.22 to 97.72] | 25.00 [0.63 to 80.59] | 25.00 [0.63 to 80.59] | 25.00 [0.63 to 80.59]
Statistical Analysis 1: Comparison: Part A & B: Double Blind Period: Placebo vs Part A: Double Blind Period: TAK-079 100 mg; Test type: Superiority; p = 0.001, Barnard's test; Risk Difference (RD) = 55.56, 95% CI 2-sided [25.11 to 81.51] — 95% CI of the difference in percentage was calculated using Miettinen-Nurminen method
Statistical Analysis 2: Comparison: Part A & B: Double Blind Period: Placebo vs Part A: Double Blind Period: TAK-079 300 mg; Test type: Superiority; p = 0.004, Barnard's test; Risk Difference (RD) = 50, 95% CI 2-sided [19.63 to 78.95] — 95% CI of the difference in percentage was calculated using Miettinen-Nurminen method
Statistical Analysis 3: Comparison: Part A & B: Double Blind Period: Placebo vs Part B: Double Blind Period: TAK-079 600 mg; Test type: Superiority; p < 0.001, Barnard's test; Risk Difference (RD) = 81.82, 95% CI 2-sided [51.24 to 94.99] — 95% CI of the difference in percentage was calculated using Miettinen-Nurminen method

4. Secondary Outcome: Percentage of Participants With Clinically Meaningful Platelet Response at Weeks 16 and 32
Description: A clinically meaningful platelet response is defined as a platelet count ≥20,000/μL above baseline on at least 2 visits without a dosing period-permitted rescue treatment in the previous 4 weeks and without any other previous rescue therapy. Percentages were rounded off to the nearest single decimal place.
Time Frame: At Weeks 16 and 32
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A & B: Double Blind Period: Placebo | Part A: Double Blind Period: TAK-079 100 mg | Part A: Double Blind Period: TAK-079 300 mg | Part B: Double Blind Period: TAK-079 600 mg | Part A: Open-label Extension (OLE) Period: TAK-079 100 mg | Part A: OLE Period: TAK-079 300 mg | Part B: OLE Period: TAK-079 600 mg
Number analyzed (Participants) | 13 | 9 | 8 | 11 | 4 | 4 | 4
percentage of participants
  Week 16 | 30.77 [9.09 to 61.43] | 66.67 [29.93 to 92.51] | 75.00 [34.91 to 96.81] | 90.91 [58.72 to 99.77] | 75.00 [19.41 to 99.37] | 50.00 [6.76 to 93.24] | 25.00 [0.63 to 80.59]
  Week 32: number analyzed (Participants) | 0 | 9 | 8 | 11 | 4 | 4 | 4
  Week 32 |  | 66.67 [29.93 to 92.51] | 75.00 [34.91 to 96.81] | 90.91 [58.72 to 99.77] | 75.00 [19.41 to 99.37] | 50.00 [6.76 to 93.24] | 25.00 [0.63 to 80.59]
Statistical Analysis 1: Comparison: Part A & B: Double Blind Period: Placebo vs Part A: Double Blind Period: TAK-079 100 mg; Test type: Superiority; p = 0.120, Barnard's test; Risk Difference (RD) = 35.9, 95% CI 2-sided [-7.22 to 67.75] — 95% CI of the difference in percentage was calculated using Miettinen-Nurminen method
Statistical Analysis 2: Comparison: Part A & B: Double Blind Period: Placebo vs Part A: Double Blind Period: TAK-079 300 mg; Test type: Superiority; p = 0.060, Barnard's test; Risk Difference (RD) = 44.23, 95% CI 2-sided [-0.83 to 73.77] — 95% CI of the difference in percentage was calculated using Miettinen-Nurminen method
Statistical Analysis 3: Comparison: Part A & B: Double Blind Period: Placebo vs Part B: Double Blind Period: TAK-079 600 mg; Test type: Superiority; p = 0.003, Barnard's test; Risk Difference (RD) = 60.14, 95% CI 2-sided [21.33 to 82.42] — 95% CI of the difference in percentage was calculated using Miettinen-Nurminen method

5. Secondary Outcome: Percentage of Participants With Hemostatic Platelet Response at Weeks 16 and 32
Description: A hemostatic platelet response is defined for participants with a baseline platelet count of <15,000/μL who achieved a platelet count of ≥30,000/μL and ≥20,000/μL above baseline on at least 2 visits without a dosing period-permitted rescue treatment in the previous 4 weeks and without any other previous rescue therapy. Percentages were rounded off to the nearest single decimal place.
Time Frame: At Weeks 16 and 32
Population: The Full Analysis Set included all randomized participants who had received at least 1 dose of study drug. Overall number of participants indicates the number of participants with data available for analyses. Number analyzed indicates the number of participants with data available for analyses at the specified time point. All participants in the 'Part A & B: Double Blind Period: Placebo' arm either transitioned to OLE Period or discontinued from the study prior to Week 32.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A & B: Double Blind Period: Placebo | Part A: Double Blind Period: TAK-079 100 mg | Part A: Double Blind Period: TAK-079 300 mg | Part B: Double Blind Period: TAK-079 600 mg | Part A: Open-label Extension (OLE) Period: TAK-079 100 mg | Part A: OLE Period: TAK-079 300 mg | Part B: OLE Period: TAK-079 600 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4 | 2 | 1 | 3
percentage of participants
  Week 16 | 0 [0.00 to 52.18] | 40.00 [5.27 to 85.34] | 25.00 [0.63 to 80.59] | 100.00 [39.76 to 100.00] | 100.00 [15.81 to 100.00] | 100.00 [2.50 to 100.00] | 0 [0.00 to 70.76]
  Week 32: number analyzed (Participants) | 0 | 5 | 4 | 4 | 2 | 1 | 3
  Week 32 |  | 40.00 [5.27 to 85.34] | 25.00 [0.63 to 80.59] | 100.00 [39.76 to 100.00] | 100.00 [15.81 to 100.00] | 100.00 [2.50 to 100.00] | 0 [0.00 to 70.76]
Statistical Analysis 1: Comparison: Part A & B: Double Blind Period: Placebo vs Part A: Double Blind Period: TAK-079 100 mg; Test type: Superiority; p = 0.187, Barnard's test; Risk Difference (RD) = 40, 95% CI 2-sided [-16.28 to 78.17] — 95% CI of the difference in percentage was calculated using Miettinen-Nurminen method
Statistical Analysis 2: Comparison: Part A & B: Double Blind Period: Placebo vs Part A: Double Blind Period: TAK-079 300 mg; Test type: Superiority; p = 0.315, Barnard's test; Risk Difference (RD) = 25, 95% CI 2-sided [-28.85 to 71.78] — 95% CI of the difference in percentage was calculated using Miettinen-Nurminen method
Statistical Analysis 3: Comparison: Part A & B: Double Blind Period: Placebo vs Part B: Double Blind Period: TAK-079 600 mg; Test type: Superiority; p = 0.004, Barnard's test; Risk Difference (RD) = 100, 95% CI 2-sided [35.12 to 100.00] — 95% CI of the difference in percentage was calculated using Miettinen-Nurminen method

ADVERSE EVENTS:
Time Frame: Up to Week 32 in each Period of the study
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Part A: Open-label Extension (OLE) Period: TAK-079 100 mg: Participants who received placebo in double-blind Part A and SFP and opted to receive treatment with TAK-079 were randomized to receive TAK-079 100 mg, SC injection, QW for 8 weeks in OLE Period of Part A. Following treatment participants were followed up for 8 weeks in a SFP and then for another 16 weeks in a LFP.
Arm/Group | Part A & B: Double Blind Period: Placebo | Part A: Double Blind Period: TAK-079 100 mg | Part A: Double Blind Period: TAK-079 300 mg | Part B: Double Blind Period: TAK-079 600 mg | Part A: Open-label Extension (OLE) Period: TAK-079 100 mg | Part A: OLE Period: TAK-079 300 mg | Part B: OLE Period: TAK-079 600 mg
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/9 | 0/8 | 0/11 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/13 | 2/9 | 0/8 | 2/11 | 1/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 9/13 | 7/9 | 5/8 | 6/11 | 2/4 | 4/4 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A & B: Double Blind Period: Placebo (N=13) | Part A: Double Blind Period: TAK-079 100 mg (N=9) | Part A: Double Blind Period: TAK-079 300 mg (N=8) | Part B: Double Blind Period: TAK-079 600 mg (N=11) | Part A: Open-label Extension (OLE) Period: TAK-079 100 mg (N=4) | Part A: OLE Period: TAK-079 300 mg (N=4) | Part B: OLE Period: TAK-079 600 mg (N=4)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A & B: Double Blind Period: Placebo (N=13) | Part A: Double Blind Period: TAK-079 100 mg (N=9) | Part A: Double Blind Period: TAK-079 300 mg (N=8) | Part B: Double Blind Period: TAK-079 600 mg (N=11) | Part A: Open-label Extension (OLE) Period: TAK-079 100 mg (N=4) | Part A: OLE Period: TAK-079 300 mg (N=4) | Part B: OLE Period: TAK-079 600 mg (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Administration site haematoma (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 2 | 0 | 1 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Essential hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site haematoma (General disorders) | 3 | 0 | 2 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0
Myopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Optic neuropathy (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post-traumatic headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT04278924/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT04278924/SAP_001.pdf